CLINICAL TRIAL: NCT02403154
Title: Prospective Randomized Comparison of Subcutaneous Internal Fixation and External Fixation for Anterior Pelvic Ring Fractures Requiring Stabilization
Brief Title: Comparison of Subcutaneous INFIX and EXFIX for Anterior Pelvic Ring Fractures Requiring Stabilization
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principle Investigator left institution
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1404651343
Record Dates: First submitted 2015-03-23; First posted 2015-03-31 (Estimated); Results first posted 2017-12-19 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-02

CONDITIONS: Anterior Pelvic Ring Fractures
Keywords: Anterior pelvic ring; Internal fixation; External fixation; Orthopaedic; Orthopedic; pubic rami
MeSH Terms: interventions — Internal Fixators; External Fixators

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Randomized to Internal Fixator (Experimental): Patient signed consent and agreed to have their treatment method randomized and the randomization system determined that their surgical intervention will be internal fixator.
  Interventions: Procedure: Internal Fixator
- Randomized to External Fixator (Experimental): Patient signed consent and agreed to have their treatment method randomized and the randomization system determined that their surgical intervention will be external fixator.
  Interventions: Procedure: External fixator
- Observational - Internal Fixator (Other): Patient signed consent but did not want to randomize their procedure and either the treating physician selected the internal fixator intervention based on their preference for the specific case or the patient chose the internal fixator.
  Interventions: Procedure: Internal Fixator
- Observational - External Fixator (Other): Patient signed consent but did not want to randomize their procedure and either the treating physician selected the external fixator intervention based on their preference for the specific case or the patient chose the external fixator.
  Interventions: Procedure: External fixator

INTERVENTIONS:
Procedure: Internal Fixator — Internal fixator refers to pins usually inserted into the iliac bones and then connected together by clamps and bars that are inserted under the skin, internally.
  Arms: Observational - Internal Fixator; Randomized to Internal Fixator
Procedure: External fixator — External fixator refers to pins usually inserted into the iliac bones and then connected together by clamps and bars that are outside of the body.
  Arms: Observational - External Fixator; Randomized to External Fixator

SUMMARY:
The purpose of this research is to compare patient outcomes of two treatment methods that are currently used as standard of care to treat anterior pelvic ring injuries that require stabilization. The two treatment methods are subcutaneous internal fixation (INFIX) and external fixation (EXFIX). Patients will be given the opportunity to opt out of randomization and participate in one of the observational arms. The first observational arm is comprised of those patients who do not want to randomize and they will undergo anterior pelvic ring stabilization according to the treating surgeon's discretion. The second observational arm will be comprised of patients who consent to be in the study but whose pelvic ring fractures do not require any form of anterior pelvic internal fixation based on the treating surgeon's opinion.

DETAILED DESCRIPTION:
The purpose of this research is to compare patient outcomes of two treatment methods that are currently used as standard of care to treat anterior pelvic ring injuries that require stabilization. The two treatment methods are subcutaneous internal fixation (INFIX) and external fixation (EXFIX). Patients will be given the opportunity to opt out of randomization and participate in one of the observational arms. The first observational arm is comprised of those patients who do not want to randomize and they will undergo anterior pelvic ring stabilization according to the treating surgeon's discretion. The second observational arm will be comprised of patients who consent to be in the study but whose pelvic ring fractures do not require any form of anterior pelvic internal fixation based on the treating surgeon's opinion. This type of injury requires follow up at 2 weeks, 6 weeks, 3 months, 6 months, 12 months, and 24 months. At each follow up appointment, the patient will be asked to complete surveys as part of the PROMIS series (Patient Reported Outcomes Measurement Information System) which will include surveys about physical function, pain, mobility, sex life satisfaction, depression, and for male patients, a survey about erectile function. In addition to the PROMIS questionnaire for pain, the investigators will also use a visual analogue pain scale and ask what the patient's satisfaction is on a scale of 0-100%. If the patient does not report to clinic for follow up, the research coordinator will call the patient to complete the study questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* One or more fractures of the anterior pelvic ring (pubic rami)
* Need for anterior pelvic ring stabilization
* Injury amenable to external as well as subcutaneous internal fixation per the treating surgeon's opinion
* Patient was ambulatory prior to sustaining the injury
* Provision of informed consent by patient or proxy

Exclusion Criteria:

* Patients with a slim build with little subcutaneous fat who cannot be treated with a subcutaneous internal fixator based on the treating surgeon's opinion
* Patients who are deemed not likely to follow-up (e.g. patients who live more than 50 miles away and patients with no fixed address)
* Moderately or severely cognitively impaired patients
* Pregnant women
* Prisoners

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zlowodzki, MD, Principal Investigator — Indiana University Health
Locations (1):
- Indiana University Health Methodist Hospital, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Arazi M, Kutlu A, Mutlu M, Yel M, Kapiciglu MI. The pelvic external fixation: the mid-term results of 41 patients treated with a newly designed fixator. Arch Orthop Trauma Surg. 2000;120(10):584-6. doi: 10.1007/s004020000142. PMID 11110141
- [Background] Gansslen A, Pohlemann T, Krettek C. [A simple supraacetabular external fixation for pelvic ring fractures]. Oper Orthop Traumatol. 2005 Sep;17(3):296-312. doi: 10.1007/s00064-005-1134-2. German. PMID 16132252
- [Background] Hupel TM, McKee MD, Waddell JP, Schemitsch EH. Primary external fixation of rotationally unstable pelvic fractures in obese patients. J Trauma. 1998 Jul;45(1):111-5. doi: 10.1097/00005373-199807000-00024. PMID 9680022
- [Background] Lindahl J, Hirvensalo E, Bostman O, Santavirta S. Failure of reduction with an external fixator in the management of injuries of the pelvic ring. Long-term evaluation of 110 patients. J Bone Joint Surg Br. 1999 Nov;81(6):955-62. doi: 10.1302/0301-620x.81b6.8571. PMID 10615965
- [Background] Majeed SA. External fixation of the injured pelvis. The functional outcome. J Bone Joint Surg Br. 1990 Jul;72(4):612-4. doi: 10.1302/0301-620X.72B4.2380212.
- [Background] Mears DC, Fu FH. Modern concepts of external skeletal fixation of the pelvis. Clin Orthop Relat Res. 1980 Sep;(151):65-72. PMID 7418325
- [Background] Tucker MC, Nork SE, Simonian PT, Routt ML Jr. Simple anterior pelvic external fixation. J Trauma. 2000 Dec;49(6):989-94. doi: 10.1097/00005373-200012000-00002. PMID 11130512
- [Background] Majeed SA. Grading the outcome of pelvic fractures. J Bone Joint Surg Br. 1989 Mar;71(2):304-6. doi: 10.1302/0301-620X.71B2.2925751.
- [Background] Riemer BL, Butterfield SL, Diamond DL, Young JC, Raves JJ, Cottington E, Kislan K. Acute mortality associated with injuries to the pelvic ring: the role of early patient mobilization and external fixation. J Trauma. 1993 Nov;35(5):671-5; discussion 676-7. doi: 10.1097/00005373-199311000-00003. PMID 8230327
- [Background] Wild JJ Jr, Hanson GW, Tullos HS. Unstable fractures of the pelvis treated by external fixation. J Bone Joint Surg Am. 1982 Sep;64(7):1010-20. PMID 7118964
- [Background] Cole PA, Gauger EM, Anavian J, Ly TV, Morgan RA, Heddings AA. Anterior pelvic external fixator versus subcutaneous internal fixator in the treatment of anterior ring pelvic fractures. J Orthop Trauma. 2012 May;26(5):269-77. doi: 10.1097/BOT.0b013e3182410577. PMID 22357081
- [Background] Gardner MJ, Mehta S, Mirza A, Ricci WM. Anterior pelvic reduction and fixation using a subcutaneous internal fixator. J Orthop Trauma. 2012 May;26(5):314-21. doi: 10.1097/BOT.0b013e318220bb22. PMID 22048189
- [Background] Merriman DJ, Ricci WM, McAndrew CM, Gardner MJ. Is application of an internal anterior pelvic fixator anatomically feasible? Clin Orthop Relat Res. 2012 Aug;470(8):2111-5. doi: 10.1007/s11999-012-2287-6. PMID 22383020
- [Background] Moazzam C, Heddings AA, Moodie P, Cole PA. Anterior pelvic subcutaneous internal fixator application: an anatomic study. J Orthop Trauma. 2012 May;26(5):263-8. doi: 10.1097/BOT.0b013e31823e6b82. PMID 22337488
- [Background] Vaidya R, Colen R, Vigdorchik J, Tonnos F, Sethi A. Treatment of unstable pelvic ring injuries with an internal anterior fixator and posterior fixation: initial clinical series. J Orthop Trauma. 2012 Jan;26(1):1-8. doi: 10.1097/BOT.0b013e318233b8a7. PMID 22048183
- [Background] Vaidya R, Kubiak EN, Bergin PF, Dombroski DG, Critchlow RJ, Sethi A, Starr AJ. Complications of anterior subcutaneous internal fixation for unstable pelvis fractures: a multicenter study. Clin Orthop Relat Res. 2012 Aug;470(8):2124-31. doi: 10.1007/s11999-011-2233-z. PMID 22219004
- [Background] Drummond M. Introducing economic and quality of life measurements into clinical studies. Ann Med. 2001 Jul;33(5):344-9. doi: 10.3109/07853890109002088. PMID 11491193
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] PELTIER LF. COMPLICATIONS ASSOCIATED WITH FRACTURES OF THE PELVIS. J Bone Joint Surg Am. 1965 Jul;47:1060-9. No abstract available. PMID 14318624
- [Background] Scaglione M, Parchi P, Digrandi G, Latessa M, Guido G. External fixation in pelvic fractures. Musculoskelet Surg. 2010 Nov;94(2):63-70. doi: 10.1007/s12306-010-0084-5. Epub 2010 Nov 18. PMID 21086087
- [Background] Pohlemann T, Bosch U, Gansslen A, Tscherne H. The Hannover experience in management of pelvic fractures. Clin Orthop Relat Res. 1994 Aug;(305):69-80. PMID 8050249
- [Background] Holstein JH, Pizanis A, Kohler D, Pohlemann T; Working Group Quality of Life After Pelvic Fractures. What are predictors for patients' quality of life after pelvic ring fractures? Clin Orthop Relat Res. 2013 Sep;471(9):2841-5. doi: 10.1007/s11999-013-2840-y. PMID 23408176
- [Background] Kabak S, Halici M, Tuncel M, Avsarogullari L, Baktir A, Basturk M. Functional outcome of open reduction and internal fixation for completely unstable pelvic ring fractures (type C): a report of 40 cases. J Orthop Trauma. 2003 Sep;17(8):555-62. doi: 10.1097/00005131-200309000-00003. PMID 14504576
- [Background] McCarthy ML, MacKenzie EJ, Bosse MJ, Copeland CE, Hash CS, Burgess AR. Functional status following orthopedic trauma in young women. J Trauma. 1995 Nov;39(5):828-36; discussion 836-7. doi: 10.1097/00005373-199511000-00005. PMID 7473997
- [Background] Mullis BH, Sagi HC. Minimum 1-year follow-up for patients with vertical shear sacroiliac joint dislocations treated with iliosacral screws: does joint ankylosis or anatomic reduction contribute to functional outcome? J Orthop Trauma. 2008 May-Jun;22(5):293-8. doi: 10.1097/BOT.0b013e31816b6b4e. PMID 18448980
- [Background] Oliver CW, Twaddle B, Agel J, Routt ML Jr. Outcome after pelvic ring fractures: evaluation using the medical outcomes short form SF-36. Injury. 1996 Nov;27(9):635-41. doi: 10.1016/s0020-1383(96)00100-3. PMID 9039360
- [Background] Suzuki T, Shindo M, Soma K, Minehara H, Nakamura K, Uchino M, Itoman M. Long-term functional outcome after unstable pelvic ring fracture. J Trauma. 2007 Oct;63(4):884-8. doi: 10.1097/01.ta.0000235888.90489.fc. PMID 18090021
- [Background] Vallier HA, Cureton BA, Schubeck D, Wang XF. Functional outcomes in women after high-energy pelvic ring injury. J Orthop Trauma. 2012 May;26(5):296-301. doi: 10.1097/BOT.0b013e318221e94e. PMID 22337480
- [Background] Lefaivre KA, Slobogean GP, Valeriote J, O'Brien PJ, Macadam SA. Reporting and interpretation of the functional outcomes after the surgical treatment of disruptions of the pelvic ring: a systematic review. J Bone Joint Surg Br. 2012 Apr;94(4):549-55. doi: 10.1302/0301-620X.94B4.27960. PMID 22434474
- [Background] Lefaivre KA, Slobogean GP, Ngai JT, Broekhuyse HM, O'Brien PJ. What outcomes are important for patients after pelvic trauma? Subjective responses and psychometric analysis of three published pelvic-specific outcome instruments. J Orthop Trauma. 2014 Jan;28(1):23-7. doi: 10.1097/BOT.0b013e3182945fe9. PMID 23571293
- [Background] Sprague S, Leece P, Bhandari M, Tornetta P 3rd, Schemitsch E, Swiontkowski MF; S.P.R.I.N.T. Investigators. Limiting loss to follow-up in a multicenter randomized trial in orthopedic surgery. Control Clin Trials. 2003 Dec;24(6):719-25. doi: 10.1016/j.cct.2003.08.012. PMID 14662277
- See also: PROMIS outcome questionnaires — http://www.nihpromis.org/software/assessmentcenter

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Randomized to Internal Fixator | Randomized to External Fixator | Observational - Internal Fixator | Observational - External Fixator
Started | 2 | 0 | 1 | 1
Completed | 0 | 0 | 0 | 0
Not Completed | 2 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized to Internal Fixator | Randomized to External Fixator | Observational - Internal Fixator | Observational - External Fixator | Total
Number analyzed (Participants) | 2 | 0 | 1 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 1 | 1 | 4
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 0 | 2
  Male | 1 | 0 | 0 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Functional Outcomes (PROMIS v1.2-Physical Function Instrument)
Description: The primary objective is to compare functional outcomes between subcutaneous internal fixation and external fixation as measured by the PROMIS v1.2-Physical Function instrument.
Time Frame: 24 hrs - 24 months
Population: No data was analyzed for this study. The PI left our institution and the study was pre-maturely closed. With such a small patient population, the data that was collected was not analyzed because achieving statistical significance was not possible.
Arm/Group | Randomized to Internal Fixator | Randomized to External Fixator | Observational - Internal Fixator | Observational - External Fixator
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Implant Breakage or Failure Rates
Description: We will compare the implant failure/breakage rate between the two interventions.
Time Frame: 24 hours - 24 months
Population: No analyses were done on this study. We did not enroll enough patients in order to come to any conclusions prior to the PI leaving the institution.
Arm/Group | Randomized to Internal Fixator | Randomized to External Fixator | Observational - Internal Fixator | Observational - External Fixator
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Infection Rates
Description: We will compare the rate of infection between the two interventions.
Time Frame: 24 hours - 24 months
Reporting Status: Not Posted

4. Secondary Outcome: Revision Surgery Rates
Description: We will compare the revision surgery rates between the two interventions.
Time Frame: 24 hours - 24 months
Reporting Status: Not Posted

5. Secondary Outcome: Health-related Qualify of Life
Description: We will ask patients multiple questionnaires to assess their quality of life after surgery. These questionnaires include: PROMIS Pain Interference, PROMIS Mobility, PROMIS Global Satisfaction with Sex Life, PROMIS Depression, Majeed score, SF-12, VAS, patient satisfaction score, and (only in men) PROMIS Erectile Function.
Time Frame: 24 hours - 24 months
Reporting Status: Not Posted

6. Secondary Outcome: Predictors of Outcome (Factors Such as Age, Gender, BMI, Additional Injuries)
Description: We will evaluate factors such as age, gender, BMI, additional injuries to see if they help predict outcome
Time Frame: 24 hours - 24 months
Reporting Status: Not Posted

7. Secondary Outcome: Compare the Functional Outcome Scores (PROMIS Pain Interference, PROMIS Mobility, PROMIS Global Satisfaction With Sex Life, PROMIS Depression, Majeed Score, SF-12, VAS, Patient Satisfaction Score, and (Only in Men) PROMIS Erectile Function)
Description: We will ask patients multiple questionnaires to asses their functional outcomes after surgery. These questionnaires include: PROMIS Pain Interference, PROMIS Mobility, PROMIS Global Satisfaction with Sex Life, PROMIS Depression, Majeed score, SF-12, VAS, patient satisfaction score, and (only in men) PROMIS Erectile Function.
Time Frame: 24 hours - 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Randomized to Internal Fixator | Randomized to External Fixator | Observational - Internal Fixator | Observational - External Fixator
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No